CLINICAL TRIAL: NCT03017027
Title: Effects of Animal Assisted Activity on Biobehavioral Stress Responses of Hospitalized Children: A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sandra M Branson, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SN-14-0202
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Psychosocial Stress
Keywords: human-animal interaction
MeSH Terms: conditions — Human-Animal Interaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapy dog visitation (TDV) (Experimental): The TDV intervention consists of a one-time 10 minute TDV with the dog handler and his/her dog interacting with the patient. The therapy dog visitation program is a currently established program and each therapy dog meets obedience, temperament, and health standards required by the organization and are deemed appropriate to therapy dog visitation. For hygienic reasons, dogs are bathed before visitation and the patient is required to wash hands before and after the visit. The TDV will be casual and not restrict the handler with conversing, which is standard practice in TDV. The therapy dog will be leashed and controlled by the dog handler. If the participant wants the dog to be placed on the bed, a clean sheet will be placed on the bed in between the dog and patient. The TDV will be casual and not restrict the handler with conversing, which is standard practice in TDV. Tactile and visual contact with the dog will be promoted.
  Interventions: Behavioral: Therapy dog visitation (TDV)
- non-TDV control (Other): Participants randomized to the control condition will receive a new plush stuffed animal for the same 10-min timeframe without any structured activities. At the end of the session, a stuffed animal will be offered to the participant to keep.
  Interventions: Behavioral: non-TDV control

INTERVENTIONS:
Behavioral: Therapy dog visitation (TDV) — The TDV intervention consists of a one-time 10 minute TDV with the dog handler and his/her dog interacting with the patient. The therapy dog visitation program is a currently established program and each therapy dog meets obedience, temperament, and health standards required by the organization and are deemed appropriate to therapy dog visitation. For hygienic reasons, dogs are bathed before visitation and the patient is required to wash hands before and after the visit. The TDV will be casual and not restrict the handler with conversing, which is standard practice in TDV. The therapy dog will be leashed and controlled by the dog handler. If the participant wants the dog to be placed on the bed, a clean sheet will be placed on the bed in between the dog and patient. The TDV will be casual and not restrict the handler with conversing, which is standard practice in TDV. Tactile and visual contact with the dog will be promoted.
  Arms: Therapy dog visitation (TDV)
Behavioral: non-TDV control — Participants randomized to the control condition will receive a new plush stuffed animal for the same 10-min timeframe without any structured activities. At the end of the session, a stuffed animal will be offered to the participant to keep.
  Arms: non-TDV control

SUMMARY:
The purpose of this study is to assess the efficacy of a 10-minute therapy dog visitation (TDV) in reducing biobehavioral stress responses among hospitalized school-age children by comparing responses between TDV and non-TDV control groups.

ELIGIBILITY:
Inclusion Criteria:

* understand English
* alert and oriented to person, place, and time
* able to complete study instruments
* able to provide saliva specimens, and
* consent from parent/legal guardian, and
* assent from child.

Exclusion Criteria:

* currently taking hormone replacement, or steroidal antiinflammatory medications
* in contact precautions at facility
* diagnosed with Addison's or Cushing's disease, and
* fears, phobias, or allergies to dogs.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety as measured by the State Anxiety Inventory for Children (STAI-C) scale | immediately before session, immediately after session
  State anxiety will be measured using the State Anxiety Inventory for Children (STAI-C), a widely used instrument with upper elementary or junior high school aged children. The instrument is composed of 20 statements that ask about how one feels at a particular moment in time with three responses from "very to not". Scores range from 20 to 80 and higher scores indicate a higher state of anxiety. Internal consistency has been demonstrated; researchers have reported acceptable reliability coefficients in hospitalized children ages 7-11 years old with Cronbach's α of .94.
Change in Positive Mood/Affect as measured by the 10-item Positive and Negative Affect Schedule for Children (10 PANAS-C) | immediately before session, immediately after session
  The 10 PANAS-C is a 10 item youth self-report measure used in child and adolescent populations which asks youth to rate adjectives of varying mood states (5 negative and 5 positive affect adjectives) on how often they feel joyful, cheerful, happy, lively, and proud and miserable, mad, afraid, scared, and sad. The item responses use a 5-point Likert scale ranging from 1 ("very slightly or none at all") to 5 ("extremely"). The 10 item PANAS-C demonstrates acceptable validity and internal consistency estimates when compared to the full-length 27-item PANAS-C scale with alpha of .86 for the positive scale; .82 for the negative scale.
Change in Negative Mood/Affect as measured by the 10-item Positive and Negative Affect Schedule for Children (10 PANAS-C) | immediately before session, immediately after session
  The 10 PANAS-C is a 10 item youth self-report measure used in child and adolescent populations which asks youth to rate adjectives of varying mood states (5 negative and 5 positive affect adjectives) on how often they feel joyful, cheerful, happy, lively, and proud and miserable, mad, afraid, scared, and sad. The item responses use a 5-point Likert scale ranging from 1 ("very slightly or none at all") to 5 ("extremely"). The 10 item PANAS-C demonstrates acceptable validity and internal consistency estimates when compared to the full-length 27-item PANAS-C scale with alpha of .86 for the positive scale; .82 for the negative scale.
Change in biological stress response as assessed by salivary cortisol levels | immediately before session, immediately after session
  Saliva samples will be collected salivary cortisol (stress), CRP, and IL-1ß (inflammatory). Time of salivary collection will be between the times of 1000-1300 to control for circadian rhythmicity. On the day of batch assay all samples will be assayed using the Salimetrics ® kits (with acceptable precision and accuracy) with an enzyme immunoassay procedure following the manufacturer's directions.
Change in biological inflammatory stress responses as assessed by salivary C-reactive protein (CRP) levels | immediately before session, immediately after session
  Saliva samples will be collected salivary cortisol (stress), CRP, and IL-1ß (inflammatory). Time of salivary collection will be between the times of 1000-1300 to control for circadian rhythmicity. On the day of batch assay all samples will be assayed using the Salimetrics ® kits (with acceptable precision and accuracy) with an enzyme immunoassay procedure following the manufacturer's directions.
Change in biological inflammatory stress responses as assessed by salivary interleukin-1beta (IL-1β) levels | immediately before session, immediately after session
  Saliva samples will be collected salivary cortisol (stress), CRP, and IL-1ß (inflammatory). Time of salivary collection will be between the times of 1000-1300 to control for circadian rhythmicity. On the day of batch assay all samples will be assayed using the Salimetrics ® kits (with acceptable precision and accuracy) with an enzyme immunoassay procedure following the manufacturer's directions.

SECONDARY OUTCOMES:
Attachment level to pets as assessed by the Pet Attitude Scale (PAS) | immediately before session
  Attachment to pets will be measured using the Pet Attitude Scale (PAS)Questionnaire.The PAS is an 18 item paper and pencil instrument with 7 Likert response statements which measures the favorableness of attitudes towards pets. Higher scores indicate more positive attitudes towards pets. Evidence of PAS-M is demonstrated with a Cronbach's alpha of .93.
Human-Animal Interaction as assessed by the Human-Animal Interaction Scale (HAIS) | immediately after session
  The Human-Animal Interaction Scale (HAIS) is a newly developed questionnaire designed to measure behavioral interactions between animal and human which predict beneficial effects to humans (Fournier, Letson, Laitalia, & Krog, 2015). The HAIS is a 26 item Likert Scale with 5 Likert response statements ranging from "not at all" to "a great deal" and is completed by the participant after the TDV.
Human-Animal Interaction as assessed by the HAIS observer questionnaire | immediately after session
  The HAIS observer questionnaire is a 24 item instrument completed by the research staff who quantifies behaviors with a percent or range in respect to the behavior observed.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M Branson, PhD, MSN, RN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States